CLINICAL TRIAL: NCT00215865
Title: HRN 003PEG-Interferon a-2b + Ribavirin for Treatment of Patients With Chronic Hepatitis C Who Have Previously Failed to Achieve a Sustained Virologic Response Following Interferon Alfa or Interferon a-2b + Ribavirin Therapy
Brief Title: PEG-Interferon a-2b + Ribavirin for Treatment of Patients With Chronic Hepatitis C Who Have Previously Failed to Achieve a Sustained Virologic Response Following Interferon Alfa or Interferon a-2b + Ribavirin Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hepatitis Resource Network (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRN 003
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Hepatitis C Virus Infection
MeSH Terms: interventions — peginterferon alfa-2b; Ribavirin

INTERVENTIONS:
Drug: PEGIntron plus ribavirin

SUMMARY:
HRN-003 STUDY SYNOPSIS

OBJECTIVE: To compare the Sustained Virologic Response (SVR) of PEGIntron plus ribavirin among patients receiving a fixed dose of PEGIntron versus weighted-adjusted dosing.

OVERVIEW OF STUDY DESIGN: This is a multi-center, randomized, open-label clinical trial using PEGIntron weight-adjusted dose by subcutaneous injection weekly + ribavirin by mouth twice daily for 48 weeks OR PEGIntron fixed dose by subcutaneous injection weekly + ribavirin by mouth twice daily for 48 weeks.

STUDY POPULATION: 600 Adult patients with chronic hepatitis C virus infection who have previously failed to achieve a sustained virologic response following interferon alfa or interferon alfa-2b plus ribavirin therapy.

DOSAGE AND ADMINISTRATION: Eligible participants will be randomized to receive PEGIntron weight-adjusted dose (1.5 mg/kg) by subcutaneous injection weekly + ribavirin 400 mg by mouth twice daily for 48 weeks OR PEGIntron fixed dose (150 mg if weight > than 80 kg or 100 mg if weight < 80 KG) by subcutaneous injection weekly + ribavirin 400 mg by mouth twice daily for 48 weeks.

EFFICACY EVALUATIONS: Laboratory analysis, quality of life assessments, and change in study medication doses will be obtained.

SAFETY EVALUATIONS: Assessment of laboratory evaluations, vital signs, incidence and severity of adverse experiences and progression of disease, as measured by HCV viral load.

STUDY DESIGN

This is a treatment protocol to evaluate the antiviral efficacy, safety and tolerability polyethylene glycol (PEG) conjugated interferon alfa-2b (PEGIntron) for the treatment of chronic hepatitis C virus infection in patients who have previously failed to achieve a sustained virologic response following interferon alfa or interferon alfa-2b plus ribavirin therapy. Patients will be stratified according to their response to the previous course of therapy (i.e. non-reponse or relapse virologic pattern

This is a multi-center, randomized, open-label clinical trial that will involve approximately 25 sites with an anticipated enrollment of 600 patients over a six-month period.

Eligible participants will be randomized to receive PEGIntron weight-adjusted dose (1.5 mg/kg) by subcutaneous injection weekly + ribavirin 400 mg by mouth twice daily for 48 weeks OR PEGIntron fixed dose (150 mg if weight > than 80 kg or 100 mg if weight < 80 KG) by subcutaneous injection weekly + ribavirin 400 mg by mouth twice daily for 48 weeks.

* Group A: PEGIntron weight -adjusted dose (1.5 mg/kg) by subcutaneous injection weekly + ribavirin 400 mg by mouth twice daily for 48 weeks (Total therapy x 48weeks).
* Group B: PEGIntron fixed dose (150 mg if weight > than 80 kg or 100 mg if weight < 80 KG) by subcutaneous injection weekly + ribavirin 400 mg by mouth twice daily for an additional 48 weeks (Total therapy x 48 weeks).

ELIGIBILITY:
Inclusion Criteria:

The patient must meet the following criteria for entry:

5.1.1 Adult male or female, age of 18 or older.

5.1.2 Serums positive for hepatitis C virus by RT-PCR or other assay (bDNA).

5.1.3 HCV genotype result must be available at screening.

5.1.4 Previous antiviral therapy with interferon or interferon plus ribavirin for at least 12 weeks with the failure to obtain a sustained virologic response.

5.1.5 No therapy with interferon alfa or interferon alfa-2b plus ribavirin or other specific anti-HCV medications within 6 weeks of the Entry visit.

5.1.6 Compensated liver disease with the following laboratory parameters at the Entry visit:

* Hemoglobin values of ³ 12 gm/dL for females or ³ 13 gm/dL for males
* WBC ³ 3,000/mm3
* Neutrophil count ³1,500/mm3
* Platelets ³ 70,000/mm3
* Prothrombin time < 2 seconds prolonged compared to control, or equivalent INR ratio
* Bilirubin within 20% of the upper limit of normal (unless non-hepatitis related factors such as Gilbert's disease explains an indirect bilirubin rise).
* Albumin > 3.0 g/dL (or within 20% of LLN)
* Serum creatinine < 1.4 mg/dL
* Hemoglobin A1C < 8.5% for diabetic patients (whether on medication and/or diet controlled)
* Thyroid Stimulating Hormone (TSH) within normal limits or thyroid disease under clinical control

5.1.7 Alpha-fetoprotein (AFP) value within normal limits obtained within the prior year. For patients with results above the upper limit of normal but < 50 ng/mL both of the following are required:

* Alpha-fetoprotein value < 50 ng/mL obtained within 3 months prior to entry AND
* Ultrasound obtained within 3 months prior to entry that is negative for evidence of hepatocellular carcinoma.

5.1.8 Reconfirmation and documentation that all sexually active female patients of childbearing potential are practicing adequate contraception (intrauterine device, oral contraceptives, progesterone implanted rods [Norplant], medroxyprogesterone acetate [Depo-Provera], surgical sterilization, barrier method [diaphragm + spermicide], or monogamous relationship with a male partner who has had a vasectomy or is using a condom + spermicide) during the treatment period and for 6 months after discontinuation of therapy. A urine pregnancy test obtained at entry prior to the initiation of treatment must be negative. Female patients must not be breast feeding. Documentation that sexually active male patients are practicing acceptable methods of contraception (vasectomy, use of a condom + spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period and for 6 months after discontinuation of therapy.

5.1.9 Anyone at high risk of coronary artery disease should have a stress test performed prior to entry. This would include, but not be limited to, patients over age 55 who have a history of ischemia or who have a significant history of hypertension, diabetes mellitus, obesity, smoking and/or strong family history of coronary artery disease. Patients with evidence of ischemia on resting or stress EKG, or a history of an arrhythmia, angina or a myocardial infarction within 12 months must be excluded.

5.1.10 Liver biopsy is not required for study entry. However, if a liver biopsy has been obtained, within three years of the initial screening visit, the pathology report will be collected with other study data.

5.1.11 Written informed consent specific for this protocol has been obtained prior to entry.

Exclusion Criteria:

The patient will be excluded from entry if any of the following criteria apply:

5.2.1 Hypersensitivity to alpha interferon or ribavirin.

5.2.2 Any other causes for chronic liver disease other than chronic hepatitis C.

5.2.3 Hemoglobinopathies (e.g., Thalassemia) or any other cause of hemolytic anemia.

5.2.4 Evidence of advanced liver disease such as a history of or presence of ascites, bleeding varices, or spontaneous encephalopathy.

5.2.5 Any known preexisting medical condition that could interfere with the patient s participation in the protocol including: CNS trauma or active seizure disorders requiring medication; poorly controlled diabetes mellitus; serious pulmonary disease; immunologically-mediated diseases; gout; or any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids.

5.2.6 Patients with evidence of ischemia on stress testing (required for patients at risk of or with a history of coronary artery disease), ECG evidence of ischemia, an arrhythmia, cardiac failure, coronary surgery, uncontrolled hypertension, angina or a myocardial infarction within 12 months.

5.2.7 Patients with clinically significant retinal abnormalities.

5.2.8 Substance abuse, such as alcohol (> 80 gm/day), I.V. drugs and inhaled drugs. If the patient has a history of substance abuse, to be considered for inclusion into the protocol, the patient must have abstained from using the abused substance for at least 1 year. Patients receiving methadone within the past year are eligible if they undergo a program of testing for substance abuse at study entry and then randomly at least every three months during therapy. Persons withdrawn from methadone therapy due to violations within their methadone program will be ineligible.

5.2.9 Patients with an alcohol consumption of > 20 gm/day are ineligible for the protocol. Patients must be counseled with regard to the need to abstain from the consumption of alcohol.

5.2.10 Concurrent use of nucleoside analogs, amantadine/rimantadine, and HIV protease inhibitors will be excluded.

5.2.11 Patients with a history of organ transplantation will be excluded.

5.2.12 Preexisting psychiatric conditions; especially depression, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or suicidal attempt are excluded. Patients with a history of mild depression may enter the protocol if they meet the following eligibility criterion and are monitored as outlined in Section 11.2 (Management of Depression During Study).

Mild depression: to include either situational depression of a limited period or depressive symptoms, which do not significantly interfere with the patients work or daily functions. Any patient with a manic element to his/her previous symptom complex will be excluded.

Detailed follow-up of each patient may be individualized according to his/her need; this would usually include further predetermined visits. Patients with a history of mild depression or patients undergoing successful treatment for mild depression will be managed as outlined in Section 11.2 (Management of Depression During Study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600

PRIMARY OUTCOMES:
1. To compare the Sustained Virologic Response (SVR) of PEGIntron plus ribavirin among patients receiving a fixed dose of PEGIntron versus weighted-adjusted dosing

SECONDARY OUTCOMES:
2. To evaluate the safety and tolerability PEG Intron in combination with ribavirin given as a fixed dose versus weight adjusted.
3. To determine the Early Virologic Response (EVR) at week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sulkowski, MD, Principal Investigator — Hepatitis Resource Network
Locations (1):
- Johns Hopkins Univesity School of Medicine, Baltimore, Maryland, United States